CLINICAL TRIAL: NCT07054736
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2 Clinical Study to Evaluate the Efficacy and Safety of XKH001 Injection in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Evaluate the Efficacy and Safety of XKH001 Injection in Patients With Moderate-to-Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Kanova Biopharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XKH001-01-II
Record Dates: First submitted 2024-12-23; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: a central randomization system will be used to randomly assign the patients to 3 dose groups of the study drug XKH001 (100 mg quaque 4 weeks , 300 mg quaque 4 weeks , 600 mg quaque 4 weeks ) and the placebo group in a 1:1:1:1 ratio, with 30 patients in each group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 100mg (Active Comparator): 100mg,quaque 4 weeks
  Interventions: Drug: XKH001 Injection; Drug: XKH001 Placebo Injection
- 300mg (Active Comparator): 300mg,quaque 4 weeks
  Interventions: Drug: XKH001 Injection; Drug: XKH001 Placebo Injection
- 600mg (Active Comparator): 600mg,quaque 4 weeks
  Interventions: Drug: XKH001 Injection; Drug: XKH001 Placebo Injection
- Placebo (Placebo Comparator): Placebo,quaque 4 weeks
  Interventions: Drug: XKH001 Placebo Injection

INTERVENTIONS:
Drug: XKH001 Injection — 100 mg quaque 4 weeks dose group: Subjects will receive 1 mL (1 vial) of XKH001 injection (100 mg) and 5 mL (5 vials) of placebo injection subcutaneously each time, once every 4 weeks, for a total of 5 times.
  300 mg quaque 4 weeks dose group: Subjects will receive 3 mL (3 vials) of XKH001 injection (300 mg) and 3 mL (3 vials) of placebo injection subcutaneously each time, once every 4 weeks, for a total of 5 times.
  600 mg quaque 4 weeks dose group: Subjects will receive 6 mL (6 vials) of XKH001 injection (600 mg) subcutaneously each time, once every 4 weeks, for a total of 5 times.
  Arms: 100mg; 300mg; 600mg
Drug: XKH001 Placebo Injection — Subjects will receive 6 mL (6 vials) of placebo injection subcutaneously each time, once every 4 weeks, for a total of 5 times.

SUMMARY:
This study will be a multicenter, randomized, double-blinded, placebo-controlled clinical study. It is planned to enroll 120 adult patients with moderate-to-severe Atopic Dermatitis whose disease cannot be adequately controlled with topical medications or for whom topical treatments are medically inadvisable.

DETAILED DESCRIPTION:
This study will be a multicenter, randomized, double-blinded, placebo-controlled clinical study. It is planned to enroll 120 adult patients with moderate-to-severe Atopic Dermatitis whose disease cannot be adequately controlled with topical medications or for whom topical treatments are medically inadvisable. With the disease severity assessed at the baseline visit-IGA: 3 points (moderate) vs. 4 points (severe) used as the stratification factors, a central randomization system will be used to randomly assign the patients to 3 dose groups of the study drug XKH001 (100 mg quaque 4 weeks , 300 mg quaque 4 weeks , 600 mg quaque 4 weeks ) and the placebo group in a 1:1:1:1 ratio, with 30 patients in each group.

This study aims to evaluate the safety, efficacy, PK and PD characteristics, and immunogenicity of XKH001 in adult patients with moderate-to-severe Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following criteria to be eligible for participation in this study:

  1. Both males and females, aged 18 to 65 years (inclusive) on the day of signing the informed consent;
  2. Diagnosed with Atopic dermatitis according to the American Academy of Dermatology consensus criteria (2014) and with a history of disease for at least 6 months prior to signing the informed consent;
  3. At the screening and baseline visits, the severity of Atopic dermatitis is classified as moderate to severe, that is, the following 4 conditions are met simultaneously; Eczema Area and Severity Index (EASI) score ≥ 16 points; Investigator's Global Assessment (IGA) score ≥ 3 points; Percent Body Surface Area (BSA) ≥10%; Weekly mean of daily Peak Pruritus Numerical Rating Scale (NRS) score ≥ 4 points;
  4. If the investigator determines that topical drug therapy used within 6 months prior to signing the informed consent was insufficiently effective or unsuitable, at least one of the following conditions must be met:

     Received ≥ 4 weeks of medium/potent topical corticosteroids (TCSs) or ≥ 2 weeks of super potent TCSs (combined with the longest treatment course recommended in the drug instructions, whichever is shorter) ± topical calcineurin inhibitors (TCIs), but did not achieve and maintain remission or a lower disease activity state (equivalent to IGA = 0 to 2); Received systemic corticosteroids (SCSs) and other systemic treatments for AD is also considered an insufficient response to topical drug therapy; Not suitable for topical drug therapy (e.g., intolerance or contraindications);
  5. Application of a stable dose of basic, mild, inactive ingredient-free topical emollients (moisturizers) twice daily for at least 7 consecutive days before the first dose and throughout the study.
  6. Subjects of childbearing potential and their partners must voluntarily use effective contraceptive methods during the study and continue for 6 months after the final dose; Note: Women of childbearing potential are those who have not undergone sterilization and either have not yet experienced menopause, have experienced menopause for less than 1 year, or have been menopausal for 1 year or more but have pathological conditions affecting menopause. Such women are considered to have potential fertility.
  7. Subjects must voluntarily sign the informed consent before any study-related procedures begin, be able to communicate effectively with the investigator, and understand and agree to adhere strictly to the protocol requirements.

Exclusion Criteria:

* Subjects who meet any of the following criteria should not be enrolled in this study:

  1. Previous treatment with biological agents for Atopic dermatitis (e.g., dupilumab, tralokinumab), XKH001, or drugs with the same target (including investigational products);
  2. Allergen-specific immunization therapy for Atopic dermatitis within 6 months prior to the first dose;
  3. Systemic drug therapy for Atopic dermatitis within 4 weeks prior to the first dose:

     Systemic corticosteroids (SCS); Immunosuppressants/immunomodulators (e.g., cyclosporin, mycophenolate mofetil, interferon-γ (IFN-γ), Janus kinase (JAK) inhibitors, azathioprine, methotrexate); Traditional Chinese medicine (including modern Chinese medicine preparations) for Atopic dermatitis treatment;
  4. Ultraviolet for Atopic dermatitis (including but not limited to narrow-band ultraviolet B (NB-UVB) and medium-to-high dose UVA1) within 4 weeks prior to the first dose;
  5. Treatment with prescription emollients or emollients containing active ingedients (e.g., ceramide, hyaluronic acid, urea, or filaggrin breakdown products) initiated during the screening period (if such emollients are used prior to signing the informed consent, they can be continued at a stable dose);
  6. ≥3 times of bleach bath therapy for Atopic dermatitis in any week within 4 weeks prior to the first dose;
  7. The following topical drug therapy for Atopic dermatitis within 2 weeks prior to the first dose:

     TCS or TCI; Other topical drugs: including but not limited to topical phosphodiesterase 4 (PDE-4) inhibitors (e.g., Crisaborole), JAK inhibitors (e.g., Ruxolitinib), traditional Chinese medicine (including modern Chinese medicine preparations);
  8. Treatment with other biological agents within 5 half-lives (if known) or 16 weeks (whichever is longer) prior to the first dose;
  9. Treatment with the investigational products (XKH001 or drugs with the same target, see Exclusion Criterion 1) or device therapy within 8 weeks or 5 half-lives (whichever is longer) prior to the first dose.
  10. Known or suspected history of immunosuppressive diseases, including history of invasive opportunistic infections (such as tuberculosis (TB), histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis), even if the infection has resolved/subsided; or abnormally frequent, recurrent, or prolonged infections as determined by the investigator (Note: Confirmed/suspected active or therapy naive latent TB must be excluded);
  11. Chronic active or acute infection requiring systemic treatment with antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks prior to the first dose; or superficial skin infection within 1 week prior to the first dose (Note: Subjects can be re-screened after the infection has resolved);
  12. Uncontrolled chronic diseases requiring extensive use of SCS, such as uncontrolled severe asthma (defined as ACQ-5 score ≥1.5 or history of ≥ 2 SCS use or hospitalization > 24 hours for asthmatic attack in the 12 months prior to signing the informed consent);
  13. Laboratory test abnormal within 7 days prior to the first dose:

      Hemoglobin (HGB) <90 g/L; Leukocyte count (WBC) <3.0×109/L; Absolute neutrophil count (ANC) <1.5×109/L; Platelet count (PLT) <90×109/L; Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN); Bilirubin total (TBIL) > 1.5 ×ULN (subjects with Gilbert syndrome >3 × ULN); Creatinine clearance (CrCl) < 50 mL/min (Cockcroft-Gault formula);
  14. Positive for hepatitis B surface antigen (HBsAg), or negative for HBsAg but positive for hepatitis B core antibody (HBcAb) and HBV-DNA > ULN, positive for antibody to hepatitis C virus (anti-HCV) and positive for HCV-RNA;
  15. History of human immunodeficiency virus (HIV) infection or positive serum HIV antibody;
  16. Other skin diseases that may interfere with the investigator's assessment during the screening period;
  17. History of neoplasm malignant within 5 years prior to signing informed consent (except for cured squamous cell carcinoma of skin in situ and basal cell carcinoma, and cured cervical carcinoma in situ);
  18. Diagnosed with active or suspected parasitic infection,, or at high risk of infection before the first administration: Unless clinical judgment (laboratory test assessment if necessary) has ruled out active infection;
  19. Combined with various serious diseases that the investigator judges may affect the patient's participation in this study, including but not limited to: Diseases that seriously affect survival, uncontrolled diabetes mellitus, ≥ Grade 2 (CTCAE 5.0) dyslipidaemia of all types (attention should be paid to excluding the influence of physiological factors such as diet), New York Heart Association (NYHA) Class 3 to 4 cardiac insufficiency, renal insufficiency requiring dialysis, Child-Pugh Class B/C liver function, demyelination diseases, active autoimmune diseases;
  20. History of mental disorder; Individuals with a history of significant mental health disorders that may affect their ability to comply with the study requirements; in addition, patients with severe anxiety or depression or suicidal ideology/behavior in the preceding 6 months will be excluded;
  21. History of alcohol abuse or various drug abuse within 2 years prior to signing informed consent;
  22. Vaccinated with attenuated live/live vaccine (including investigational vaccines) within 12 weeks prior to the first administration, or planning to be vaccinated with attenuated live/live vaccine during the study;
  23. Major surgery (craniotomy, thoracotomy, laparotomy, etc.) within 4 weeks prior to the first administration, or planning to undergo major surgery during the study;
  24. Within 2 weeks prior to the first administration, there is severe blood loss (total blood volume ≥ 500 mL), or received blood products, hematopoietic growth factors (e.g. granulocyte colony-stimulating factor G-CSF), albumin infusion;
  25. Women who are known to be pregnant or have childbearing potential have a positive serum human chorionic gonadotropin (HCG) test at screening, or are breastfeeding, or are planning to become pregnant or breastfeed during the study;
  26. Subjects with known allergy to the study drug, any ingredient in the study drug formulation, or history of allergy to protein drugs;
  27. Other conditions that the investigator considers unsuitable for participation in this study;
  28. Subjects who are currently enrolled in another clinical trial or investigational study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective1 | Week16
  Proportion of subjects with an Investigator's Global Assessment (IGA) score of 0 or 1 (clear or almost clear) and a reduction of ≥2 points from baseline to Week 16.
Primary Objective2 | Week16
  Proportion of subjects with Treatment Emergent Serious Adverse Events (TESAEs) from baseline to Week 16

SECONDARY OUTCOMES:
Secondary Objective1 | Week16
  Proportion of subjects with improvement (Reduction ≥4 Points) of Pruritus Numerical Rating Scale (NRS) Score from baseline to Week 16
Secondary Objective2 | Week16
  Percent change from baseline in Peak Daily Pruritus Numerical Rating Scale (NRS) Score to Week 16
Secondary Objective3 | Week4
  Proportion of subjects with improvement (Reduction
  ≥4 Points) of Pruritus Numerical Rating Scale (NRS) Score from baseline to Week 4
Secondary Objective4 | Weeks 4, 8, 12, 16, 20, 24, and 28;
  Change from baseline in percent Body Surface Area (BSA) affected at Weeks 4, 8, 12, 16, 20, 24, and 28;
Secondary Objective5 | Weeks 4, 8, 12, 16, 20, 24, and 28;
  Percent change from baseline in IGA 0/1 and reduction of ≥ 2, mean EASI score and weekly average of peak daily Pruritus Numeric Rating Scale (NRS) at Weeks 4, 8, 12, 16, 20, 24, and 28;
Secondary Objective6 | weeks 4, 8, 12, 16, 20, 24
  Percent change in AD specific symptomatic and quality of life (QOL) assessment with AD control tool (ADCT) from baseline to weeks 4, 8, 12, 16, 20, 24

OTHER OUTCOMES:
Exploratory Objective | Week16
  The correlation between the expression levels of skin tissue biomarkers (including: IL-25 and its signaling pathway-related proteins in skin tissue) and clinical efficacy will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Dr, Principal Investigator — Peking University People's Hospital
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No